CLINICAL TRIAL: NCT00086177
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Efficacy, Safety, and Tolerability of 8% Progesterone Vaginal Gel in Preventing Preterm Delivery in Pregnant Women at Increased-Risk for Preterm Delivery
Brief Title: Vaginal Progesterone to Reduce the Risk of Another Preterm Birth
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juniper Pharmaceuticals, Inc. (Industry)
Responsible Party: George W. Creasy, MD, FACOG, VP Clinical Research, Columbia Laboratories
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: COL-1620-300
Record Dates: First submitted 2004-06-25; First posted 2004-06-29 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Pregnancy
Keywords: Pregnancy,; prevention of preterm birth,; prevention of preterm labor,
MeSH Terms: interventions — Progesterone; Crinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Progesterone 8% vaginal gel
  Interventions: Drug: 8% progesterone vaginal gel
- 2 (Placebo Comparator): Placebo Vaginal Gel
  Interventions: Drug: Placebo Vaginal Gel

INTERVENTIONS:
Drug: 8% progesterone vaginal gel — Progesterone 8% Vaginal gel, once daily, maximum duration from 18 07 weeks gestation to 37 0/7 weeks gestation
  Other Names: Prochieve; Crinone
  Arms: 1
Drug: Placebo Vaginal Gel — Placebo vaginal gel, once daily, maximum duration from 18 07 weeks gestation to 37 0/7 weeks gestation
  Arms: 2

SUMMARY:
This research study is being conducted at over 12 pregnancy research centers in the US. The study will compare an investigational treatment with a placebo (a treatment without medication). Neither the investigators nor the patients in the trial will know which treatment has been assigned. All study medications will be given vaginally once a day. Treatment will begin before pregnancy week 23 and will continue until the end of pregnancy week 36.

DETAILED DESCRIPTION:
Patients who participate are to have:

* A single baby pregnancy (no twins or triplets allowed)
* Patients will start treatment before pregnancy week 23
* Patients must have a previous preterm birth (a "preemie")
* Patients must be 18-45 years of age

ELIGIBILITY:
Inclusion Criteria:

1. The subject has a history of a documented spontaneous singleton preterm delivery (hospital or clinic record, letter from healthcare provider, or birth certificate) from 20 0/7 to 35 0/7 weeks gestational age with the immediate preceding pregnancy or has a cervical length of 2.5 cm or less measured by transvaginal ultrasound with the current pregnancy. "Spontaneous preterm delivery" is a delivery (<35 weeks), either vaginal or cesarean, that is initiated by either preterm PROM followed by contractions or preterm labor initiated with in-tact membranes. A previous preterm delivery secondary to an incompetent cervix where a cerclage is considered for this pregnancy is not considered a preterm delivery (please see Exclusion Criteria No. 10). Subjects enrolled based on a history of preterm delivery may have had a pregnancy loss (or losses) at <20 0/7 weeks gestational age between the preceding preterm delivery and the current pregnancy.
2. The female subject is between 18 and 45 years of age at the time of screening.
3. The pregnancy has an estimated gestational age between 16 0/7 weeks and 22 6/7 weeks.
4. The subject speaks either English or a common local language.
5. The subject has voluntarily signed the Informed Consent Form and associated forms after having the contents explained, and all her questions are answered to her satisfaction and understanding.
6. In the opinion of the investigator, the subject is able to understand the study and is able to give informed consent, as well as participate in it and adhere to study procedures.

Exclusion Criteria:

1. The subject has a previous history of an adverse reaction to progesterone or any component present in Prochieve® 8% vaginal gel.
2. The subject has been treated with a progestogen within the previous 4 weeks.
3. The subject is currently being treated for a seizure disorder, has an unstable psychiatric disorder, is taking antihypertensive therapy for chronic hypertension at the time of enrollment, has a history of congestive heart failure or chronic renal failure, or has uncontrolled diabetes mellitus (known end-organ dysfunction secondary to vascular disease).
4. The subject has active thrombophlebitis or a thromboembolic disorder, or a history of hormone-associated thrombophlebitis or thromboembolic disorders.
5. The subject has liver dysfunction or disease.
6. The subject has known or suspected malignancy of the breast or genital organs.
7. The subject is currently participating in another investigational study or has participated in an investigational drug study within one month prior to screening for this study.
8. The subject's current pregnancy is complicated by a major fetal anomaly or known chromosomal abnormality.
9. The subject has a uterine anatomic malformation (bicornuate uterus, septate uterus)
10. The subject has a multifetal gestation.
11. The subject has a cervical cerclage in place or has plans to have one placed during the current pregnancy.
12. The subject, in the judgment of the investigator, will be unable or unwilling to comply with study-related assessments and procedures.
13. The subject currently has preterm rupture of membranes, vaginal bleeding, known or suspected amnionitis, or signs or symptoms of preterm labor at the time of enrollment.
14. The subject is HIV positive with a CD4 count of _<350 cells/mm3 and is receiving more than 1 medication to prevent the transfer of AIDS to the fetus.
15. The subject has placenta previa or a low-lying placenta. The subject will be considered for the study if she is not at risk for increased bleeding and has not been given any vaginal precautions.
16. The subject's qualifying preterm delivery was an indicated delivery without preterm labor (i.e. delivery performed for fetal distress, maternal eclampsia/preeclampsia, fetal death, or amnionitis in the absence of contractions).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 636 (Actual)
Dates: Start 2004-04; Primary Completion 2007-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Frequency of delivery <=32 weeks | 18 weeks gestation through delivery

SECONDARY OUTCOMES:
Frequency of delivery preterm | 18 weeks gestation through delivery
Response to tocolytic therapy | Onset of preterm labor through resolution or delivery
Number of infant hospital days from delivery to discharge | Delivery date through hospital discharge date of infant

CONTACTS AND LOCATIONS:
Overall Officials: George W Creasy, MD, Study Director — VP Clinical Research; Columbia Laboratories, Inc
Locations (45):
- United States (45):
  - University of South Alabama Department of OBGYN, Mobile, Alabama
  - Visions Clinical Research-Tucson, Tucson, Arizona
  - Women's Health Department, Colton, California
  - SanDiego Perinatal Center, San Diego, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Kaiser Permanente, Denver, Colorado
  - Northside Maternal Fetal Specialists, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Illinois, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Maternal Fetal Medicine Norton Suburban Hospital, Louisville, Kentucky
  - Maternal Fetal Medicine &Woman's Health Research, Baton Rouge, Louisiana
  - Louisiana State University Health Sciences Center-Shreveport, Shreveport, Louisiana
  - Johns Hopkins Community Physicians, Baltimore, Maryland
  - Holy Cross Hospital, Silver Springs, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center -MFM, Brighton, Massachusetts
  - St. Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Department of OBGYN, St. Barnabas Medical Center, Livingston, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - St. Luke's - Roosevelt Hospital, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Pitt County Memorial Hospital, Greenville, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - Ohio Permanente Medical Group, Bedford, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - MacDonald Clinical Trials Unit, University Hospitals of Cleveland, Cleveland, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University Medical Center, Philadelphia, Pennsylvania
  - Abington Primary Women's Healthcare, Willow Grove, Pennsylvania
  - University Medical Group, Dept of OB/GYN, Greenville, South Carolina
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - Gynecology & Obstetrics, Memphis, Tennessee
  - Womens Partner In Health, Austin, Texas
  - Health Central Women's Care, Dallas, Texas
  - Clinical Research Center of Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Texas Tech Health Sciences Center - Odessa, Odessa, Texas
  - EVMS Maternal-Fetal Medicine, Hofheimer Hall, Norfolk, Virginia
  - West Virginia University, Morgantown, West Virginia

REFERENCES:
- [Background] da Fonseca EB, Bittar RE, Carvalho MH, Zugaib M. Prophylactic administration of progesterone by vaginal suppository to reduce the incidence of spontaneous preterm birth in women at increased risk: a randomized placebo-controlled double-blind study. Am J Obstet Gynecol. 2003 Feb;188(2):419-24. doi: 10.1067/mob.2003.41. PMID 12592250
- [Result] O'Brien JM, Adair CD, Lewis DF, Hall DR, Defranco EA, Fusey S, Soma-Pillay P, Porter K, How H, Schackis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Progesterone vaginal gel for the reduction of recurrent preterm birth: primary results from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):687-96. doi: 10.1002/uog.5158. PMID 17899572
- [Result] DeFranco EA, O'Brien JM, Adair CD, Lewis DF, Hall DR, Fusey S, Soma-Pillay P, Porter K, How H, Schakis R, Eller D, Trivedi Y, Vanburen G, Khandelwal M, Trofatter K, Vidyadhari D, Vijayaraghavan J, Weeks J, Dattel B, Newton E, Chazotte C, Valenzuela G, Calda P, Bsharat M, Creasy GW. Vaginal progesterone is associated with a decrease in risk for early preterm birth and improved neonatal outcome in women with a short cervix: a secondary analysis from a randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2007 Oct;30(5):697-705. doi: 10.1002/uog.5159. PMID 17899571
- [Derived] O'Brien JM, Defranco EA, Adair CD, Lewis DF, Hall DR, How H, Bsharat M, Creasy GW; Progesterone Vaginal Gel Study Group. Effect of progesterone on cervical shortening in women at risk for preterm birth: secondary analysis from a multinational, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2009 Dec;34(6):653-9. doi: 10.1002/uog.7338. PMID 19918965